CLINICAL TRIAL: NCT05420662
Title: The Effects of Vaginal Manipulator Use on the Residual Vaginal Length and Operative Outcomes in Abdominal Hysterectomy Operations
Brief Title: The Application of Vaginal Manipulator in Abdominal Hysterectomy Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Şener Gezer, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KAEK /05.bI.05
Record Dates: First submitted 2022-06-12; First posted 2022-06-15 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Abdominal Hysterectomy
Keywords: Vaginal Manipulator

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal Manipulator Group (Experimental): In this group of patients, abdominal hysterectomy surgery will be performed with the vaginal manipulator. After cutting and suturing uterine arteries, cardinal and sacrouterine ligaments are preserved by using a vaginal manipulator. The manipulator applied vaginally prevents unnecessary vaginal length loss by ensuring that the vaginal cuff is cut from the top point of the vagina.
  Interventions: Procedure: Manipulation of vagina during abdominal hysterectomy operation
- Classical Abdominal Hysterectomy Group (Active Comparator): In this group of patients, abdominal hysterectomy surgery will be performed in a conventional way, by cutting the cardinal and sacrouterine ligaments.
  Interventions: Procedure: Classical conventional abdominal hysterectomy operation

INTERVENTIONS:
Procedure: Manipulation of vagina during abdominal hysterectomy operation — The manipulator applied vaginally prevents unnecessary vaginal length loss by ensuring that the vaginal cuff is cut from the top point.
  Arms: Vaginal Manipulator Group
Procedure: Classical conventional abdominal hysterectomy operation — Classical conventional abdominal hysterectomy operation without any manipulation from the vagina.
  Arms: Classical Abdominal Hysterectomy Group

SUMMARY:
If a vaginal manipulator is used for abdominal hysterectomy, the vagina can be cut and separated from the cervix without cutting the Cardinal and Sacrouterine ligaments and protecting the top of the vaginal tissue (Portio vaginalis). In this way, both the shortening of the vagina and the prolapse of the vaginal cuff can be prevented. In addition, the duration of hysterectomy surgery is significantly shortened.

DETAILED DESCRIPTION:
In a classical abdominal hysterectomy, the Cardinal ligaments and the Sacrouterine ligaments are cut before the uterus leaves the vagina, and the vaginal cuff is cut deeper in the vagina over the cervix and separated from the vagina. During this procedure, the vaginal tissue in the Portio vaginalis comes out and causes a loss of vaginal length. If a vaginal manipulator is used for abdominal hysterectomy, the vagina can be cut and separated from the cervix without cutting the Cardinal and Sacrouterine ligaments and protecting the top of the vaginal tissue (Portio vaginalis). In this way, both the shortening of the vagina and the prolapse of the vaginal cuff can be prevented. In addition, the duration of hysterectomy surgery is significantly shortened.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent hysterectomy due to abnormal uterine bleeding
* Myoma uteri, little than 5 cm which does not disrupt the uterine anatomy

Exclusion Criteria:

* Myoma uteri, which disrupts the uterine anatomy
* Intra-abdominal adhesions
* Endometrial intraepithelial neoplasia
* Endometrial cancer
* Ovarian cancer
* Cervical cancer

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Vaginal Length Difference | Preoperative one hour and postoperative one hour
  The difference between preoperative and postoperative vaginal length will be calculated

SECONDARY OUTCOMES:
Operation time | One to two hours
  Skin-to-skin operation time and the time frame from the beginning of the hysterectomy to the moment when the uterus leaves the vagina.

CONTACTS AND LOCATIONS:
Overall Officials: Şener Gezer, MD, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kiyak H, Karacan T, Ozyurek ES, Turkgeldi LS, Kadirogullari P, Seckin KD. Abdominal Hysterectomy with a Uterine Manipulator Minimizes Vaginal Shortening: A Randomized Controlled Trial. J Invest Surg. 2021 Oct;34(10):1052-1058. doi: 10.1080/08941939.2020.1744774. Epub 2020 Apr 2. PMID 32238020